CLINICAL TRIAL: NCT03423043
Title: Comparison of Low Dose Computed Tomography to Conventional Dose Computed Tomography in the Evaluation of Distal Radius Fractures
Brief Title: Low Dose CT Distal Radius Fractures
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00089089
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-06

CONDITIONS: Radius Fractures
MeSH Terms: conditions — Radius Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Distal Radius Fracture Patients: Adult patients who have sustained a Distal Radius Fracture.
  Interventions: Radiation: Low Dose CT Scan of the Wrist

INTERVENTIONS:
Radiation: Low Dose CT Scan of the Wrist — A low dose CT scan will be obtained in patients with a distal radius fracture of the wrist.

SUMMARY:
This study is a prospective, departmental funded study examining the outcomes of Low Dose CT scans compared to Conventional Dose CT scans in patients who present to Duke University with a Distal Radius Fracture.

DETAILED DESCRIPTION:
The purpose of this study is to compare the use of a conventional dose computed tomography scan (C-CT) to a low dose computed tomography scan (L-CT) in the assessment of articular displacement, and development of a treatment plan for intraarticular distal radius fractures in an effort to reduce the radiation exposure to future patients with this injury pattern. Reviewers will be tasked with reporting data aimed at investigating 3 primary outcome measures: 1) Are L-CT images of sufficient quality to be used for diagnostic purposes, 2) Can accurate measurements of step and gap displacement be made on L-CT images, 3) Do proposed treatment plans change with the use of L-CT relative to those chosen based on C-CT images We hypothesize that reviewers will find L-CT images of sufficient image quality for diagnostic purposes, measurements of step and gap displacement will not be significantly different between L-CT and C-CT, and no significant differences in treatment options will be chosen based on the use of L-CT rather than C-CT for the same fracture. The secondary aim will be to evaluate the interobserver and intraobserver reliability of L-CT in evaluating intraarticular fractures of the distal radius.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be age 18 years or older.
* Subject must have sustained an intraarticular distal radius fracture which undergo closed reduction and application of a below-elbow splint.
* Subjects whos injury occurred less than 2 weeks prior to the time of enrollment.

Exclusion Criteria:

* Subject is under the age of 18 years.
* Subject is unable to speak English for completion of consent process.
* Subject sustained pathologic fracture.
* Subject sustained open fracture.
* Subject is a pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet above eligibility criteria who present to the Duke University Medical Center for distal radius fracture evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Low Dose CT Images of Sufficient Diagnostic Quality | 12 months.
  Low Dose CT Images will be compared to a standard dose to assess image quality.

SECONDARY OUTCOMES:
Step Displacement | 12 months
  Representative CT images will be used to measure the step displacement of each fracture.
Gap Displacement | 12 months
  Representative CT images will be used to measure the gap displacement of each fracture.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data is not planned to be shared outside of the collaborators of this project within the Duke University Medical Center. The data will only be reviewed by the study personnel listed on the Institutional Review Board (IRB), and not intended to be shared with an external institution or industry.
  However, when submitting data for manuscripts and publication purposes, all data will be deidentified of any public health information. All Protected Health Information (PHI) will be kept in a locked cabinet in the PI's office at Duke University and/or in a protected/encrypted folder in a file separate from the study information. Data will be analyzed by study team members using a computer that is password protected, and stored securely in encrypted Duke servers. Study files will be backed up onto Dr. Klifto's folder in a secure server provided to faculty in the Department of Orthopaedic Surgery. The subjects will not be identified in any reports or publications from this study.

REFERENCES:
- [Background] Karl JW, Olson PR, Rosenwasser MP. The Epidemiology of Upper Extremity Fractures in the United States, 2009. J Orthop Trauma. 2015 Aug;29(8):e242-4. doi: 10.1097/BOT.0000000000000312. PMID 25714441
- [Background] Knirk JL, Jupiter JB. Intra-articular fractures of the distal end of the radius in young adults. J Bone Joint Surg Am. 1986 Jun;68(5):647-59. PMID 3722221
- [Background] Tanabe K, Nakajima T, Sogo E, Denno K, Horiki M, Nakagawa R. Intra-articular fractures of the distal radius evaluated by computed tomography. J Hand Surg Am. 2011 Nov;36(11):1798-803. doi: 10.1016/j.jhsa.2011.08.021. Epub 2011 Oct 5. PMID 21981830
- [Background] Arora S, Grover SB, Batra S, Sharma VK. Comparative evaluation of postreduction intra-articular distal radial fractures by radiographs and multidetector computed tomography. J Bone Joint Surg Am. 2010 Nov 3;92(15):2523-32. doi: 10.2106/JBJS.I.01617. PMID 21048172
- [Background] das Gracas Nascimento V, da Costa AC, Falcochio DF, Lanzarin LD, Checchia SL, Chakkour I. Computed tomography's influence on the classifications and treatment of the distal radius fractures. Hand (N Y). 2015 Dec;10(4):663-9. doi: 10.1007/s11552-015-9773-8. Epub 2015 Jun 4. PMID 26568720
- [Background] Katz MA, Beredjiklian PK, Bozentka DJ, Steinberg DR. Computed tomography scanning of intra-articular distal radius fractures: does it influence treatment? J Hand Surg Am. 2001 May;26(3):415-21. doi: 10.1053/jhsu.2001.22930a. PMID 11418901
- [Background] Mettler FA Jr, Huda W, Yoshizumi TT, Mahesh M. Effective doses in radiology and diagnostic nuclear medicine: a catalog. Radiology. 2008 Jul;248(1):254-63. doi: 10.1148/radiol.2481071451. PMID 18566177
- [Background] Griffey RT, Sodickson A. Cumulative radiation exposure and cancer risk estimates in emergency department patients undergoing repeat or multiple CT. AJR Am J Roentgenol. 2009 Apr;192(4):887-92. doi: 10.2214/AJR.08.1351. PMID 19304691
- [Background] Sodickson A, Baeyens PF, Andriole KP, Prevedello LM, Nawfel RD, Hanson R, Khorasani R. Recurrent CT, cumulative radiation exposure, and associated radiation-induced cancer risks from CT of adults. Radiology. 2009 Apr;251(1):175-84. doi: 10.1148/radiol.2511081296. PMID 19332852
- [Background] Konda SR, Goch AM, Leucht P, Christiano A, Gyftopoulos S, Yoeli G, Egol KA. The use of ultra-low-dose CT scans for the evaluation of limb fractures: is the reduced effective dose using ct in orthopaedic injury (REDUCTION) protocol effective? Bone Joint J. 2016 Dec;98-B(12):1668-1673. doi: 10.1302/0301-620X.98B12.BJJ-2016-0336.R1. PMID 27909130
- [Background] Konda SR, Howard DO, Gyftopoulos S, Davidovitch RI, Egol KA. Computed tomography scan to detect intra-articular air in the knee joint: a cadaver study to define a low radiation dose imaging protocol. J Orthop Trauma. 2013 Sep;27(9):505-8. doi: 10.1097/BOT.0b013e3182821505. PMID 23287769
- [Background] Cole RJ, Bindra RR, Evanoff BA, Gilula LA, Yamaguchi K, Gelberman RH. Radiographic evaluation of osseous displacement following intra-articular fractures of the distal radius: reliability of plain radiography versus computed tomography. J Hand Surg Am. 1997 Sep;22(5):792-800. doi: 10.1016/s0363-5023(97)80071-8. PMID 9330135